CLINICAL TRIAL: NCT03239236
Title: Modified Rapid Sequence Induction in Morbidly Obese Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding available
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thomas Hamp, Univ. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Modified RSI in morbidly obese
Record Dates: First submitted 2017-06-16; First posted 2017-08-04 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Anesthesia Intubation Complication
MeSH Terms: interventions — Anesthetics; Blood Gas Analysis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- t-RSI (Experimental): Rapid sequence induction t-RSI. Traditional rapid sequence induction with Anesthetics. Preoxygenation via face mask, no ventilation with no PEEP until intubation. Aspiration of gastric air via nasogastric tube at the beginning of laparoscopy. Impression of gastric inflation at laparoscopy will be assessed by taking images of the stomach at the beginning of laparoscopy.
  Arterial blood gas samples will be taken at different time points.
  Interventions: Procedure: Rapid sequence induction t-RSI; Drug: Anesthetics; Diagnostic Test: Aspiration of gastric air via nasogastric tube; Diagnostic Test: Impression of gastric inflation at laparoscopy.; Diagnostic Test: Arterial blood gas
- m-RSI-PEEP (Experimental): Rapid sequence induction m-RSI-PEEP. Modified rapid sequence induction with Anesthetics and PEEP. Preoxygenation via facemask with PEEP of 10 mbar. PEEP will be continued until intubation.
  Aspiration of gastric air via nasogastric tube at the beginning of laparoscopy. Impression of gastric inflation at laparoscopy will be assessed by taking images of the stomach at the beginning of laparoscopy.
  Arterial blood gas samples will be taken at different time points.
  Interventions: Procedure: Rapid sequence induction m-RSI-PEEP; Drug: Anesthetics; Diagnostic Test: Aspiration of gastric air via nasogastric tube; Diagnostic Test: Impression of gastric inflation at laparoscopy.; Diagnostic Test: Arterial blood gas
- m-RSI-vent (Experimental): Rapid sequence induction m-RSI-vent. Modified rapid sequence induction with Anesthetics and intermittent ventilation. Preoxygenation via facemask with 10 mbar PEEP and 8 mbar pressure support. Backup frequency set at 10/min. Ventilation via anesthetic machine until intubation.
  Aspiration of gastric air via nasogastric tube at the beginning of laparoscopy. Impression of gastric inflation at laparoscopy will be assessed by taking images of the stomach at the beginning of laparoscopy.
  Arterial blood gas samples will be taken at different time points.
  Interventions: Procedure: Rapid sequence induction m-RSI-vent; Drug: Anesthetics; Diagnostic Test: Aspiration of gastric air via nasogastric tube; Diagnostic Test: Impression of gastric inflation at laparoscopy.; Diagnostic Test: Arterial blood gas
- m-RSI-vent-cric (Experimental): Rapid sequence induction m-RSI-vent-cric. Modified rapid sequence induction with Anesthetics and intermittent ventilation and cricoid pressure. Same as "modified rapid sequence induction with intermittent ventilation" arm with additional cricoid pressure.
  Aspiration of gastric air via nasogastric tube at the beginning of laparoscopy. Impression of gastric inflation at laparoscopy will be assessed by taking images of the stomach at the beginning of laparoscopy.
  Arterial blood gas samples will be taken at different time points.
  Interventions: Procedure: m-RSI-vent-cric; Procedure: Cricoid Pressure; Drug: Anesthetics; Diagnostic Test: Aspiration of gastric air via nasogastric tube; Diagnostic Test: Impression of gastric inflation at laparoscopy.; Diagnostic Test: Arterial blood gas

INTERVENTIONS:
Procedure: Rapid sequence induction t-RSI — Preoxygenation via face mask, no ventilation with no PEEP until intubation
  Arms: t-RSI
Procedure: Rapid sequence induction m-RSI-PEEP — Preoxygenation via facemask with PEEP of 10 mbar. PEEP will be continued until intubation.
  Arms: m-RSI-PEEP
Procedure: Rapid sequence induction m-RSI-vent — Preoxygenation via facemask with 10 mbar PEEP and 8 mbar pressure support. Backup frequency set at 10/min. Ventilation via anesthetic machine until intubation.
  Arms: m-RSI-vent
Procedure: m-RSI-vent-cric — Preoxygenation via facemask with 10 mbar PEEP and 8 mbar pressure support. Backup frequency set at 10/min. Ventilation via anesthetic machine until intubation.
  Arms: m-RSI-vent-cric
Procedure: Cricoid Pressure — Cricoid Pressure will be applied during RSI until laryngoscopy
  Arms: m-RSI-vent-cric
Drug: Anesthetics — Induction agents will be administered as quick boluses (Propofol 2,5mg/kg total body weight, max 350mg, Fentanyl 250mcg, Rocuronium 1,2mg/kg ideal body weight).
  Other Names: Induction Agents
Diagnostic Test: Aspiration of gastric air via nasogastric tube — A nasogastric tube will be inserted at the beginning of laparoscopy and the air from the stomach will be aspirated with a syringe. The amount of air will be measured in ml.
Diagnostic Test: Impression of gastric inflation at laparoscopy. — The impression of gastric inflation at laparoscopy. At the beginning of laparoscopy, images of the stomach will be recorded.
Diagnostic Test: Arterial blood gas — Arterial blood gases will we drawn at different time points to investigate oxygenation during the procedure. Blood gases will be taken before pre-oxygenation, before anesthesia induction, before laryngoscopy, immediately after intubation when the cuff of the tracheal tube is inflated.

SUMMARY:
This study investigates the effect of 4 different methods of rapid sequence induction (RSI) in morbidly obese patients on the amount of air insufflation into the stomach.

DETAILED DESCRIPTION:
100 adult patients with a body mass index > 40 undergoing elective laparoscopic surgery will be included. Patients with a history of previous bariatric surgery or with an anticipated difficult airway will be excluded.

The randomization will be 1:1:1:1 stratified for gastro-esophageal reflux disease.

All groups will receive standardized preoperative continuous positive airway pressure (CPAP) therapy.

In the operation theater, Group one will receive pre-oxygenation for 3 minutes via a tight fitting face mask without positive end-expiratory pressure (PEEP). Induction agents will be administered as quick boluses (Propofol 2,5mg/kg total body weight, max 350mg, Fentanyl 250mcg, Rocuronium 1,2mg/kg ideal body weight) and tracheal intubation will be performed after 1 minute. No bag mask ventilation will be performed in-between.

Group 2 will receive pre-oxygenation via a tight face mask with a PEEP of 10 mbar for 3 minutes. The same induction agents as in group one will be administered. PEEP via facemask will be continued for one minute and tracheal intubation will be performed.

Group 3 will receive pre-oxygenation via a tight fitting facemask with a PEEP of 10 mbar with additional pressure support of 8 mbar and a back up ventilation frequency will be set to 10/min. After the same induction agents are given as in group 1, patients will receive non-invasive ventilation via ventilator at the settings described earlier for group 3.

Group 4 will receive the same induction as group 3, in addition a cricoid pressure will be applied during the non invasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40
* American Society of Anesthesiology Class 1-3
* Elective laparoscopic surgery

Exclusion Criteria:

* Pregnant or breastfeeding patients
* Previous bariatric surgery
* Anticipated difficult airway

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Amount of air aspirated with a gastric tube | at the beginning of the laparoscopy
  The amount of air that can be aspirated via a nasogastric tube at the beginning of laparoscopy. A nasogastric tube will be inserted at the beginning of laparoscopy and the air from the stomach will be aspirated with a syringe. The amount of air will be measured in ml.

SECONDARY OUTCOMES:
Gastric inflation | at the beginning of laparoscopy
  The impression of gastric inflation at laparoscopy. At the beginning of laparoscopy, images of the stomach will be recorded. These images will afterwards be reviewed in a blinded fashion by three different investigators. The investigators will rate their impression of gastric inflation (empty, mildly inflated, inflated, very inflated).
partial pressure of oxygen in arterial blood (paO2) | before pre oxygenation, before anesthesia induction, before laryngoscopy, immediately after intubation when the cuff of the tracheal tube is inflated
  Arterial blood gases will we drawn at different time points to investigate oxygenation during the procedure. Blood gases will be taken before pre-oxygenation, before anesthesia induction, before laryngoscopy, after intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Plöchl, Professor, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided